CLINICAL TRIAL: NCT03567941
Title: A Randomized, Double-Blind, Double-Dummy, Active- and Placebo-Controlled, 4-Way Crossover Study to Evaluate the Relative Abuse Potential of Hydrocodone Bitartrate and Acetaminophen 6 × 10/325 mg Tablets Compared to NORCO® 6 × 10/325 mg Tablets and Placebo in Non-Dependent, Recreational Opioid Users When Administered Orally Under Fed and Fasted Conditions
Brief Title: To Evaluate the Relative Abuse Potential of Hydrocodone Bitartrate and Acetaminophen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLR_16_07
Record Dates: First submitted 2018-03-20; First posted 2018-06-26 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Single dose
  Interventions: Drug: Placebo; Drug: Hydrocodon bitartrate-acetaminophen arm 1; Drug: Hydrocodon bitartrate-acetaminophen arm 2; Drug: Reference
- Hydrocodon bitartrate-acetaminophen arm 1 (Experimental): Single dose
  Interventions: Drug: Placebo; Drug: Hydrocodon bitartrate-acetaminophen arm 1; Drug: Hydrocodon bitartrate-acetaminophen arm 2; Drug: Reference
- Hydrocodon bitartrate-acetaminophen arm 2 (Experimental): Single dose
  Interventions: Drug: Placebo; Drug: Hydrocodon bitartrate-acetaminophen arm 1; Drug: Hydrocodon bitartrate-acetaminophen arm 2; Drug: Reference
- Reference (Active Comparator): Single dose
  Interventions: Drug: Placebo; Drug: Hydrocodon bitartrate-acetaminophen arm 1; Drug: Hydrocodon bitartrate-acetaminophen arm 2; Drug: Reference

INTERVENTIONS:
Drug: Placebo — Tablet orally administered under fasting
Drug: Hydrocodon bitartrate-acetaminophen arm 1 — Tablet orally administered under fasted conditions
Drug: Hydrocodon bitartrate-acetaminophen arm 2 — Tablet orally administered under fed conditions
Drug: Reference — Tablet orally administered under fasted conditions

SUMMARY:
Evaluation of abuse potential in recreational abusers of Hydrocodone Bitartrate and Acetaminophen versus NORCO®.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects 18 to 55 years of age.
2. Opioid users who have used opioids for recreational purposes and or is an avid opioid user.

Exclusion Criteria:

1. Substance or alcohol dependence (excluding nicotine and caffeine) within the past 2 years.
2. Heavy smoker and/or is unable to abstain from smoking or unable to abstain from the use of prohibited nicotine containing products for at least 6 hours during the in-clinic periods.
3. Difficulty swallowing large number of pills.
4. Subjects who have had a tattoo or body piercing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Drug Liking | 15 weeks
  Visual analog scale on score from 0 to 100

CONTACTS AND LOCATIONS:
Locations (1):
- SPARC Site 1, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No